CLINICAL TRIAL: NCT05859685
Title: Efficacy of Manual Ankle Therapy on Fear of Falls, Range of Motion, and Functionality and Stability in Geriatric Patients. A Randomized, Double-blind Clinical Study
Brief Title: Manual Ankle Therapy on Fear of Falls, Range of Motion, and Functionality and Stability in Geriatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Rubén Cuesta-Barriuso, PhD, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RoM-Ankle
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2023-05

CONDITIONS: Old Age; Atrophy
MeSH Terms: conditions — Atrophy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: All evaluations will be carried out by one evaluator, blinded to the study conditions and the assignment of the players to the two study groups.
  The patients included in the control group underwent the same techniques as those indicated for the experimental group, but without sliding or placing joint tension. The periodicity and administration times will be the same.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The patients included in the experimental group will undergo the following manual therapy techniques:
  * Talar dorsal sliding technique. A dorsal mobilization of the talus will be performed, with the patient in the supine position and dorsiflexion of the ankle, without pain or discomfort. The physiotherapist will exercise an anteroposterior mobilization of the talus, with a dorsal glide
  * Mulligan movement mobilization technique: The patient will be in a standing position, with the ankle to be treated forward. You will be given an aid or support in the upper extremity to maintain stability.
  Interventions: Other: Experimental
- Control group (Placebo Comparator): The patients included in the control group underwent the same techniques as those indicated for the experimental group, but without sliding or placing joint tension. The periodicity and times of administration will be the same
  Interventions: Other: Control

INTERVENTIONS:
Other: Experimental — Manual therapy techniques:
  * Talar dorsal sliding technique. Dorsal mobilization of the talus, with the patient in the supine position and ankle dorsiflexion, without pain or discomfort. The physiotherapist will exercise an anteroposterior mobilization of the talus, with a dorsal glide
  * Mulligan movement mobilization technique: The patient will be in a standing position, with the ankle to be treated forward. You will be given an aid or support in the upper extremity to maintain stability.
  Arms: Experimental group
Other: Control — The patients included in the control group underwent the same techniques as those indicated for the experimental group, but without sliding or placing joint tension. The periodicity and times of administration will be the same
  Arms: Control group

SUMMARY:
The range of movement of the ankle decreases with age and the plantar arch decreases, adopting a more pronated position of the foot.

The main objective is to analyze the effectiveness of manual therapy using ankle joint techniques in geriatric patients.

Randomized, double-blind clinical trial with follow-up period. Subjects will be assigned to control and experimental groups using a data analysis tool (Excel).

The dependent variable will be the fear of falls. The secondary variables will be the range of movement in dorsiflexion of the ankle, and the functionality and stability of the lower limbs.

Three evaluations will be carried out. A baseline measurement before the start of the study (T0), after the intervention (T1) and after a 3-week follow-up period (T2).

A manual therapy protocol will be carried out, lasting 3 weeks with 1 weekly session. Each session will last 10 minutes. The patients included in the experimental group will undergo the following manual therapy techniques: talus dorsal sliding technique and joint technique in "8" on the Lisfranc and Chopart joints. The patients included in the control group underwent the same techniques as those indicated for the experimental group, but without sliding or placing joint tension. The periodicity and times of administration will be the same

ELIGIBILITY:
Inclusion Criteria:

* Subjects older than 65 years
* Subjects of both sexes
* With impaired balance and gait
* With joint limitation of ankle dorsiflexion
* With established functionality or stability deficits (for example, who need third parties or technical aids to walk (crutches))

Exclusion Criteria:

* People with cognitive impairment that prevents their collaboration in the intervention and the different evaluations
* People with inability to stand
* People who have not given their written consent.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-05-06 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline fear of falls after treatment and at 3 three weeks | Screening visit, within the first seven days after treatment and after three weeks follow-up
  With the Short Falls Efficacy Scale-International, the confidence and ability of a person to avoid a fall while performing basic activities of daily living will be evaluated. The Spanish version of this instrument has shown high reliability (α>0.87). It consists of 7 items with a score of 7 to 28 points (higher scores indicate less confidence and ability).

SECONDARY OUTCOMES:
Change from baseline ankle range of motion after treatment and at 3 three weeks | Screening visit, within the first seven days after treatment and after three weeks follow-up
  The range of movement of the ankle will be measured with a goniometer, following the protocol of Martin et al. The axis will be placed at the lower vertex of the lateral malleolus, the fixed arm parallel to the longitudinal midline of the leg and the mobile arm parallel to the longitudinal midline of the fifth metatarsal. This instrument has shown high reliability (ICCC=0.8-0.9). The higher the graduation, the greater range of motion
Change from baseline biomechanical analysis of gait and balance after treatment and at 3 three weeks | Screening visit, within the first seven days after treatment and after three weeks follow-up
  It will be evaluated with an Rs Scan® pressure platform and FootScan® pressure measurement system. This device measures plantar pressure using an X-Y array of resistive pressure sensitive sensors that are sequentially scanned. The system records pressure data when the subject is standing or walking on the platform. The measurements will be made with the basic platform of 0.5m with 4096 sensors with resistive technology and 300Hz data acquisition frequency. The biomechanics of gait will be analyzed with the analysis of the probes and the static balance in a time of 30 seconds.
Change from baseline functionality after treatment and at 3 three weeks | Screening visit, within the first seven days after treatment and after three weeks follow-up
  The 2-Minutes Walking Test (2MWT) will be used. It will be carried out in a closed corridor, with a length of 30 m delimited between cones. Before the test, participants must rest for at least 10 minutes. Subsequently, they will be told that they must walk the circuit around the cones as fast as possible, but without running, for 2 minutes. They will be allowed to use aids to walk, slow down or stop to rest if necessary. The distance traveled at the end of the 2 minutes will be recorded by the evaluator. This instrument has shown excellent test-retest reliability (ICC = 0.97)

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Study Director — Universidad de Oviedo
Locations (1):
- Universidad Católica San Antonio de Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided